CLINICAL TRIAL: NCT02183662
Title: Safety and Pharmacokinetics of Single Rising Oral Doses of BI 224436 ZW at 6.2 mg, 12.5 mg, 25 mg, 50 mg, 100 mg, 200 mg, 400 mg, 600 mg, 900 mg and 1200 mg Dose Levels in Healthy Male Volunteers (Randomized, Double-blind, Placebo-controlled Within Dose Groups)
Brief Title: Safety and Pharmacokinetics of Single Rising Oral Doses of BI 224436 ZW in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1277.1
Record Dates: First submitted 2014-07-07; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BI 224436 (Experimental)
  Interventions: Drug: BI 224436
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo to BI 224436

INTERVENTIONS:
Drug: BI 224436
  Arms: BI 224436
Drug: Placebo to BI 224436
  Arms: Placebo

SUMMARY:
To investigate safety and pharmacokinetics of BI 224436 ZW

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Age ≥21 and Age ≤50 years
3. Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and the local legislation.

Exclusion Criteria:

1. Any finding of the medical examination (including blood pressure (BP), pulse rate (PR) and electrocardiogram (ECG)) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. HIV infection and other chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within one month prior to administration or during the trial
12. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
13. Inability to refrain from smoking on trial days
14. Alcohol abuse (more than 60 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the treatment period)
18. Any laboratory value outside the reference range that is of clinical relevance
19. A baseline prolongation of QT/QTc interval (e.g., a QTc interval ≥450 ms)
20. A history of additional risk factors for Torsades de points (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
21. Bradycardia (PR <60 beats/min)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
maximum measured concentration of the analyte in plasma | up to 72 hours
area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to 24 | up to 24 hours

SECONDARY OUTCOMES:
area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity | up to 72 hours
minimum observed concentration at 24 hours | up to 24 hours
terminal half-life of the analyte in plasma | up to 72 hours
time from dosing to maximum measured concentration of the analyte in plasma | up to 72 hours
apparent clearance of the analyte in plasma | up to 72 hours
apparent volume of distribution during the terminal phase λz | up to 72 hours
apparent volume of distribution | up to 72 hours
mean residence time of the analyte in the body after single oral administration | up to 72 hours
terminal rate constant in plasma | up to 72 hours
the last measurable concentration in the concentration-time profile | up to 72 hours
the extrapolated Area under the curve from the time of the last measurable concentration in the concentration-time profile to infinity | up to 72 hours
the percentage of the Area under the concentration-time curve until infinity, that is determined by extrapolation | up to 72 hours
amount of analyte that is eliminated in urine from the time point t0 to time point t4 | up to 4 hours
amount of analyte that is eliminated in urine from the time point t4 to time point t8 | from 4 to 8 hours
amount of analyte that is eliminated in urine from the time point t8 to time point t12 | from 8 to 12 hours
amount of analyte that is eliminated in urine from the time point t12 to time point t24 | from 12 to 24 hours
fraction of analyte eliminated in urine from time point t0 to time point t24 | up to 24 hours
renal clearance of the analyte from the time point t0 until the time point t24 | up to 24 hours